CLINICAL TRIAL: NCT03043131
Title: Comparative Analysis Between Ringer's Lactate vs Acetate Containing Balanced Crystalloid Solution (Plasma Lyte-A) as Cardiopulmonary Bypass Prime
Brief Title: Comparative Analysis Between Ringer's Lactate vs Plasma Lyte-A as Cardiopulmonary Bypass Prime
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Doniparthi Pradeep, Junior Resident, Department of General Surgery, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NK/2997/MS/603
Record Dates: First submitted 2016-11-26; First posted 2017-02-03 (Estimated); Last update posted 2017-02-03 (Estimated); Status verified 2017-02

CONDITIONS: Cardiopulmonary Bypass
Keywords: Cardiopulmonary bypass prime; Plasma Lyte - A; Ringer;s lactate; Acidosis
MeSH Terms: conditions — Acidosis | interventions — Plasmalyte A; Ringer's Lactate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ringer Lactate (Active Comparator): patients randomized to this arm are given ringer's lactate solution for cardiopulmonary bypass prime, which is the standard practice
  Interventions: Drug: Ringer Lactate
- Plasmalyte A (Experimental): patients randomized to this arm are given Plasma Lyte - A solution for cardiopulmonary bypass prime
  Interventions: Drug: Plasmalyte A

INTERVENTIONS:
Drug: Plasmalyte A — Plasma Lyte -A is administered intra operatively to maintain the hemodynamic status of patients
  Other Names: Acetate containing balanced crystalloid solution
  Arms: Plasmalyte A
Drug: Ringer Lactate — Ringer's lactate is administered intra operatively to maintain the hemodynamic status of patients
  Other Names: RL
  Arms: Ringer Lactate

SUMMARY:
Metabolic acidosis is a frequent problem in cardiopulmonary bypass. The cause is poorly understood, but it appears to be multifactorial. It is assumed to be result of hypoperfusion with resultant lactatemia. And other theories include bicarbonate dilution to excessive proton activity and diluting fluid.The main three contributors for the development of metabolic acidosis are stress of anaesthesia, surgery and Cardio Pulmonary Bypass(CPB) prime.Even after research discussion and debate, there is no agreement upon ideal prime.The literature is extensive, comparing different types of colloids, colloids versus crystalloids, synthetic versus organic, and inclusion of numerous additions in an attempt to make a grossly unphysiological state the least disruptive to the body as possible

DETAILED DESCRIPTION:
REVIEW OF LITERATURE The ideal prime for Cardiopulmonary Bypass (CPB) has never been fully established. The development of acid-base disorders during some routine cases and the possible contribution to this from priming fluids caused this hospital to question its protocol.

Plasma Lyte-A injection, pH 7.4, is a sterile, nonpyrogenic isotonic solution, for intravenous administration. Each 100mL contains 368mg of Sodium acetate Trihydrate, (C2H3NaO2.3H2O), 502 mg of Sodium gluconate (C6H11NaO7), 526 mg of sodium chloride, (NaCl), 30 mg of Magnesium chloride (MgCl2.6H2O) ,37 mg of Potassium chloride, (KCl). It contains no anti microbial agents. pH is adjusted with sodium hydroxide. Its pH is 7.4 (6.5 to 8).

One litre has an ionic concentration of 27mEq of acetate, and 23mEq of gluconate, 5mEq of potassium, 140mEq sodium, 3mEq of magnesium, 98mEq of chloride. The osmolarity of 294mOsm/ml. Normal physiological osmolarity range is 280 to 310mOsm/lit. Administration of substantially hypertonic solutions may cause vein damage. The calorie content is 21 k.Cal/lit.

100ml of Ringer's lactate contains 320mg of sodium lactate, 600mg of sodium chloride, 40mg of potassium chloride, and 27mg of calcium chloride. It is equivalent to sodium of 130mEq, calcium of 3mEq, potassium of 4mEq, bicarbonate of 28mEq and chloride of 109mEq. Hence it has value as source of water, electrolytes and calories.

Infusion fluids that do not contain the physiological buffer base bicarbonate tend to produce dilutional acidosis because infusion of such solution dilutes (reduces) the HCO3- concentration (buffer base) of the entire extracellular compartment, while the partial pressure of CO2 (buffer acid) remains constant. Dilution may be isovolemic (normovolemic), i.e., HCO3- is lost along with the blood and the blood or extracellular fluid volume is restored to normal with a solution that is free of HCO3-, or the ECFV is expanded with a bicarbonate-free solution to produce hypervolemia. A decrease in arterial pH to 7.20 was observed in a dog model after infusion of 1,500mL of 0.9 % NaCl solution in 5 minutes, while no such effect was observed in dogs infused with the same volume of a solution containing 30mmol/L of NaHCO3. In summary, dilutional acidosis is predictable and defined as an iatrogenic disruption brought on by bicarbonate dilution in the entire extracellular space which may be associated with hyperchloremia or hypochloremia depending on whether dilution was produced by infusion of a hyperchloremic or hypochloremic solution.

Dilutional acidosis can be prevented by the use of adequate concentrations of metabolizable anions to replace HCO3-.The following anions of organic acids, acetate (acetic acid), lactate (lactic acid), gluconate (gluconicacid), malate or hydrogen malate (malic acid), and citrate (citric acid) may be used as metabolizable bases. Consuming H+ ions and oxygen in the process, these anions are metabolized in the intact liver (mainly lactate) or in muscle (mainly acetate and malate) to produce HCO3-. At pH 7.40, carbonic acid (H2CO3) is the only H+ ion source of the body (while supplied at a low concentration of 1.2mmol/L, H2CO3 can be synthesized freely from CO2 + H2O). HCO3- is therefore released in equimolar amounts. For every mole of acetate, gluconate, or lactate oxidized, one mole of bicarbonate is produced, while for every mole of malate or citrate oxidized, 2 or 3 moles of bicarbonate are produced, respectively. The two latter metabolizable anions would thus produce excessively high, unphysiological bicarbonate concentrations. If an infusion fluid contains metabolizable anions in concentrations exceeding the lack of bicarbonate, infusion-induced alkalosis is a likely consequence, called rebound alkalosis. Metabolic alkalosis is always iatrogenic. The normal plasma acetate concentration is very low and has been reported to range from 0.06 to 0.2mmol/L. Patients undergoing acetate hemodialysis have had plasma acetate levels as high as 6.5mmol/L.

Acetate Metabolism

Any metabolic pathway must be electro-neutral on balance. Acetate (the base the patient is infused with) is therefore oxidized in the form of acetic acid (after taking up H+). Two moles of O2 are required per mole of acetic acid. The chemical equation for the reaction of sodium acetate with oxygen is:

CH3-COONa + 2 O2<------> CO2 + H2O + NaHCO3

Two important conclusions can be drawn from this equation:

1. For every mole of acetate oxidized, one mole of bicarbonate is produced; this is the expected effect of acetate for HCO3- replacement or alkalization.
2. For every two moles of O2 consumed, only one mole of CO2 is produced. This is a surprising "side" effect in that the respiratory quotient (RQ) for acetate is only 0.5. Compared with glucose (dextrose), which has a RQ of 1.0, this means that the metabolism of acetate causes only half the inhaled O2 to be exhaled as CO2.

Compared with HCO3-, acetate has practically the same effect Lactate Metabolism CH3-CH-COONa + 3 O2 <----->CO2 + 2H2O + 2NaOH CO2 +H2O <----->H2CO3 H2CO3 + NaOH<---->NaHCO3+H2O Summary : Na lactate +3O2 <-----> 2CO2+2 H2O+NaHCO3 At the basal metabolic rate (BMR), the myocardium, muscle, brain, intestinal mucosa, and red blood cells produce approximately 1mmol of lactate/kg/h, and more than half of it is eliminated by the liver.

At the BMR, gluconeogenesis accounts for approximately 20 % and oxidation for approximately 80 % of lactate metabolism. When lactate is supplied exogenously, up to 70 % of lactate can be used as a substrate for gluconeogenesis. Intrahepatic gluconeogenesis ceases once pH falls below 7.1, or a base excess (BE) of -15mmol/L. Incipient hepatic dysfunction (increases in bilirubin and SGOT) quickly results in lactate concentrations as high as 8mmol/L, which are associated with very high mortality. Compared with acetate, lactate infusion is characterized by a relatively slow onset of alkalization and, therefore, has been called "delayed HCO3- infusion". Peak lactate turnover has been reported to be approximately 450mmol/h. As glucose levels may increase quite significantly after lactate administration, it comes as no surprise that intra-operatively administered Ringer's lactate may cause glucose concentrations to double in diabetics. Plasma lactate has similarly high predictive power to base excess for mortality in patients with various forms of shock including cardiac, hemorrhagic, and septic shock. Subsequent mortality is approximately 50 % when plasma lactate (not blood lactate) exceeds 4 to 7mmol/L in the first 24 to 48 hours of shock. An initial value of only 3mmol/L plasma lactate concentration predicts a 25 % mortality of cardiac, hemorrhagic, and septic shock patients.

Many physicians apparently are not aware that the use of lactate-containing infusion fluids (such as Ringer's lactate) or blood products (such as packed red cells) and the diagnostic use of lactate as a marker of hypoxia are mutually exclusive.

Lilley A et al conducted a survey to analyze practice of CPB circuit priming. The response rate was 74%. It was found that no two units in the UK used the same prime. The most common reason for fluid choice was historical beliefs and there appeared to be little perceived association between prime and acidosis on bypass. The results revealed that there is no consensus in the UK of the preferential prime for CPB, suggesting the effect this aspect has is not fully understood.

Liskaser FJ et al studied role of pump prime in the etiology and pathogenesis of CPB acidosis and reported that fluid with no lactate significantly limits the increase in the serum lactate concentrations in post operative period. In this study he has compared the Ringer's solution and Plasma Lyte-A. He has done a prospective, double blind randomized trial, which was conducted in a tertiary health care centre with 22 patients, undergoing CPB for coronary artery bypass surgery. He concluded that CPB induced metabolic acidosis appears to be iatrogenic in nature and derived from effect of pump prime fluid on acid-base balance. The extent of such acidosis and its duration varies according the type of pump prime.

Hayhoe M et al conducted a study and concluded that in patients receiving pump prime rich in chloride and polygeline, metabolic acidosis in CPB is mainly due to iatrogenic chloride concentration and unmeasured strong anions.Sampling of arterial blood at four time intervals: post-induction, on CPB during cooling and rewarming, and at skin closure. Measurement of serum Na+ K+, Mg++ ,Ca++, Cl-, bicarbonate, and phosphate concentrations, arterial blood gases, and serum albumin, lactate, and pyruvate concentrations at each collection point. Analysis of findings according to quantitative physicochemical principles, including calculation of the strong ion difference apparent, the strong ion difference effective, and the strong ion gap (SIG). All patients developed a mild metabolic acidosis. The median serum standard bicarbonate concentration decreased from 25.0mEq/l post-induction to 22.3mEq/l at cooling and 22.2mEq/l at rewarming (p < 0.05).The standard base excess decreased from a median of 1.55mEq/l prior to CPB, to ±2.50mEq/l at cooling,±1.65mEq/l at rewarming and,±0.85mEq/l at skin closure(p <0.001). This mild metabolic acidosis occurred despite a decrease in the median serum lactate concentration from 3.20mEq/l post-induction to 1.83, 1.80, and 1.58mEq/l at the three other time points. The increase in the median serum chloride concentration from 104.9mEq/l post induction to111.0,111.1,and110.0mEq/l at the subsequent time points (p<0.0001) was the main cause of the acidosis. There was also a significant increase in the SIG of 3.8mEq/l at cooling and rewarming (p<0.0001), suggesting a role for other unmeasured anions (polygeline) in the genesis of this acidosis. He has concluded that using quantitative biophysical methods, it can be demonstrated that, in patients receiving a pump prime rich in chloride and polygeline, the metabolic acidosis of CPB is mostly due to iatrogenic increases in serum chloride concentration and unmeasured strong anions (SIG). Its development is partially attenuated by iatrogenic hypoalbuminaemia. Changes in lactate concentrations did not play a role in the development of metabolic acidosis in the patients.

Himpe D et al conducted a study by adding lactate to prime fluid during CPB and concluded that exogenous lactate attenuated the CPB related acidosis. He has conducted study on twenty patients scheduled for coronary surgery was studied prospectively. All patients were treated identically, except for the prime, which either contained lactate or was lactate free. Just before bypass and before coming off bypass, haemoglobin, glucose, plasma osmolality and colloid osmotic pressure were determined; albumin, lactate, sodium, potassium, ionized calcium, magnesium, phosphate, arterial pH, pCO2, bicarbonate, and base excess were measured for use in Stewart's analysis. Metabolic acidosis had resolved by the end of bypass with the lactated prime. Although the strong ion gap (apparent minus effective strong ion difference) increased significantly in both groups, its composition differed significantly between the groups. The Stewart technique detected polyanionic gelatin as a weak acid component contributing to the unidentified anion fraction. Colloid osmotic pressure was maintained in both groups. He concluded that exogenous lactate attenuates acidosis related to CPB.

Weinberg LD et al conducted a randomized blinded study of 50 adult patients undergoing elective Coronary Artery Bypass Graft or heart valve replacement. Both groups received a prime solution of 2000mL; anions lactate and chloride (Hartmann's), or anions acetate, gluconate and chloride (Plasma Lyte-A).Blood was collected immediately prior to CPB (BL), 2-minutes (T2), 5-minutes (T5), 10-minutes (T10), 30-minutes (T30), and 60-minutes (T60) on CPB. Patient characteristics were evenly matched. On delivery of pump prime both groups developed metabolic acidosis. Plasma Lyte-A, standard BE: 0.53mmol/L (BL) to -3.03mmol/L (T2), P<0.001; Hartmann's standard BE: 0.42mmol/L (BL) to -2.20mmol/L (T2), P<0.001. There was a surge in the Plasma Lyte-A group's SIG - 1.39mEq/L (BL) to 12.13mEq/L (T2), P<0.001, remaining elevated at T60 (6.22mEq/L). The SIG in the Hartmann's group increased from 0.43mEq/L (BL) to 2.00mEq/L (T2). The Hartmann's group experienced a significant lactate surge at 2 minutes (P<0.001) remaining elevated at T60; there was no hyperlactatemia in the Plasma Lyte-A group. There was significant hyperchloraemia with Hartmann's compared to Plasma Lyte-A. He concluded that the mechanism of acidosis with Hartmann's solution was due to combination of iatrogenic hyperlactatemia and hyperchloraemia. The mechanism with Plasma Lyte-A was a production of unmeasured anions (likely acetate and gluconate). Metabolic acidosis can be treated or minimized by widening the strong ion difference (alkalinizing effect), maintaining a higher sodium concentration (use of sodium bicarbonate), while decreasing the chloride through use of intravenous fluids with lower chloride concentrations compared the Hartmann's solution and Plasma Lyte-A.

Morgan TJ et al designed a bicarbonate based crystalloid based circuit balanced on physio-chemical principles with a strong ion difference of 24mEq/l compared its acid base effects with those of Plasma-Lyte 148 a multiple electrolyte replacement solution containing acetate and gluconate (total 50mEq/l). Twenty patients with normal acid base status undergoing elective cardiac study were randomized 1:1 to a 2 litres prime of either bicarbonate based fluid or Plasma-Lyte 148. With the trial fluid metabolic acid base status was normal following cardiopulmonary bypass initiation (standard base excess 0.1 (1.3) mEq/l, mean, SD), whereas plasma Lyte - 148 produced a slight metabolic acidosis (standard base excess 2.2 (2.1)mEq/l, mean, SD). Estimated group difference after baseline adjustment was 3.6mEq/l (95% confidence interval 2.1 to 5.1 p=0.0001). By late bypass mean standard base excess in both groups was normal (0.8(2.2)mEq/l Vs -0.8 (1.3) p=0.5). Strong ion gap values were unaltered with trial fluid, but with the Plasma Lyte - 148 increased significantly on bypass initiation. (15.2(2.5)mEq/l Vs 2.5(1.5)mEq p<0.0001 )remaining elevated in late bypass. (8.4(3.4)mEq/l Vs5.8(2.4)mEq/l p<0.05). They have concluded that bicarbonate based crystalloid with strong ion difference of 24mEq/l is balanced for cardiopulmonary bypass in patients with normal acid base status, whereas Plasma-Lyte 148 trigger a surge of unmeasured anions, persisting throughout the bypass. These are likely to be acetate and gluconate.

Alston RP et al studied the effects of changing the solutions back to Hartmann's on metabolic acidosis that develops during CPB in patients undergoing heart surgery. He has taken two groups of patients were studied. The first received Ringer's (n = 63) and the second Hartmann's solution (n = 66). Arterial blood samples were taken before induction of anaesthesia and towards the end of CPB. Samples were analyzed in a blood gas analyzer. Results: Hydrogen ion concentration increased from 38 (4) to 41 (7)mmol/L in the Ringer's group, but decreased from 38 (5) to 36 (6)mmol L-1 in the Hartmann's group. Changes in PaCO2 (0.77, p < 0.001) and volume of fluid administered (r = 0.23, p < 0.01) were significant univariate correlates of change in hydrogen ion concentration, but haemoglobin concentration was not (r < 0.01, p = 0.97). Analysis of variance for repeated measures found significant difference between subject effects on the change in hydrogen ion concentration during CPB caused by the choice of intravascular solution used (p < 0.001) and PaCO2 (p = 0.001), but not as a result of the volume of solution administered (p > 0.10). He concluded that changing the solutions used for priming and intravascular volume replacement from Ringer's to Hartmann's was associated with a reduction in metabolic acidosis that developed during CPB.

Murray DM et at al conducted a study to define the true incidence and nature of acidosis in paediatric patients post cardiac surgery. In their study Tissue acidosis occurred overall in 60 of 150 samples. This was due to raised unmeasured acids alone in 44 of 60 (73.3%), raised lactate alone in six of 60 (10%), and a combination of the two in ten of 60 (16.6%). Hyperchloremia occurred in 19 of 150 samples overall and 12 of 25 (48%) samples immediately after cardiopulmonary bypass. Measured base deficit showed a poor correlation with true tissue acidosis (p < 0.001) and the worst discriminatory ability. They concluded that metabolic acidosis occurs frequently post cardiac surgery and is largely due to raised unmeasured acids and less commonly raised lactate. Hyperchloremia is common, particularly after cardiopulmonary bypass.

AIMS AND OBJECTIVES Primary Objective To study whether Ringer's lactate and Plasma Lyte-A, as CPB circuit prime, are similar in terms of changes in acid base status in perioperative period of patients undergoing cardiac surgery Secondary Objective When used as cardiopulmonary bypass prime, effect of Plasma Lyte-A and Ringer's lactate on renal parameters

1. Urea
2. Creatinine
3. Creatinine clearance

MATERIALS AND METHODS Type of study: A single centre prospective comparative randomized, double blinded, controlled study Study design Between July 2016 and September 2017, a total of 60 patients who fit the inclusion criteria, undergoing normothermic cardiopulmonary bypass for Coronary Artery Bypass Graft and heart valve surgeries, in cardiothoracic and vascular surgery department of Postgraduate Institute of Medical Education and Research, Chandigarh will be recruited into the study. Full informed consent will be obtained from each eligible patient before enrolment into the study. Demographic and patient data will be recorded during recruitment.

Baseline evaluation will be carried out before inclusion and include:

1. Medical history including any comorbidities or prior surgical intervention
2. Physical examination
3. Routine Laboratory tests including: Haemogram, Liver function tests, Renal function tests, Coagulogram.
4. Base line arterial blood gases with lactate
5. 2D echo cardiogram Patients will be divided into two groups. Group R will be given Ringer lactate as CPB prime and Group P will be given Plasma Lyte-A as CPB prime. Haemoglobin level will be maintained at8gm/dl on CPB and 10gm/dl before separation from bypass. At the end the parameters of the study will be compared between the two groups.

The following data will be recorded for all the patients:

1. Arterial blood gases (ABG) before induction
2. ABG five minutes after CPB
3. ABG at the end of the termination of CPB
4. ABG after half an hour stay in the ICU soon after the patient is shifted from completion of surgery
5. ABG before the patient is extubated.
6. Additives and their amounts added to the prime to correct acidosis
7. Intra operative aortic cross clamp time
8. Duration of bypass
9. Post operative investigations haemogram, liver function tests, renal function tests and coagulogram at interval of 12 hours, 24 hours and 48 hours.

4. DATA COLLECTION AND FOLLOW UP: In this study, Patients will be divided into two groups. Each Patient will be allotted either of the groups by a computer generated random number using the software link http://graphpad.com/quickcalcs/randomize2/. The arterial blood gases along with lactate levels are recorded at the time of induction, and followed, five minutes after CPB, at the end of the termination of CPB, half an hour stay in the ICU soon after the patient is shifted from completion of surgery and at the time of extubation. Urea levels, Creatinine levels and Creatinine clearance will be recorded pre operatively and will be followed in immediate post-operative period and 12 hours after surgery, 24 hours surgery, and 48 hours after surgery.

STASTISTICAL ANALYSIS As discussed in methodology, the primary objective is to compare Plasma Lyte-A and Ringer's lactate as cardiopulmonary bypass prime on the basis of ABG.

Hence the lactate is primary outcome variable which is quantitative in nature. It is presumed that the variable lactate will follow normal distribution and therefore, the appropriate statistical test to study the significant difference at each condition between the two groups will be independent t-test.

If it doesn't follow normal distribution non-parametric alternative of independent t-test will be used like Mann-Whitney U-test.

To see the trend within the group at different time intervals, repeated measure ANOVA will be used.

Summary statistics for the quantitative variables will be represented by mean, SD and for the qualitative variable will be represented by number or percentage.

To see the trend, line chart will be used. All the proposed tests will be used at 5% level of significance (α) All the statistical computation will be done on Statistical Package for Social Sciences software (SPSS version 22.0) on windows operating system.

ETHICAL JUSTIFICATION Recent studies have demonstrated that better outcomes in terms of acidosis with the use of Plasma Lyte-A (Acetate containing balanced crystalloid solution) as Cardiopulmonary Bypass prime, being more physiological to plasma in composition. Thus, the present study compares the effects of Plasma Lyte-A as a priming fluid with respect to ringer lactate.

According to the guidelines set up by Indian Council of Medical Research (1994) and Helsinki Declaration (modified 2000), the following will be adhered to in all patients enrolled in the study.

1. The patients involved in the research project will be volunteers and informed participants.
2. Each patient will be adequately informed of the aims, methods, sources of funding, any possible conflicts of interest, institutional affiliations of the researcher, the anticipated benefits and potential risks of the study and the discomfort it may entail to him/her and the remedies thereof.
3. Every precaution will be taken to respect the privacy of the patient, the confidentiality of the patients information and to minimize the impact of the study on his/her physical and rental integrity and his/her personality.
4. The patient will be given the right to abstain from participation in the study or to with draw consent to participate at any time of the study without reprisal.
5. Due care and caution will be taken at all stages of the research to ensure that the patient is put to the minimum risk, suffer from no irreversible adverse effects and, generally, benefit from and by the research or experiment. There will be no risk to the patient as a simple investigation like complete haemogram, arterial blood gas analysis is routinely done for all patients undergoing treatment.
6. Written informed consent will be obtained from all the patients included in the study.

   PARTICIPANT INFORMATION SHEET INVESTIGATOR: DR. DONIPARTHI PRADEEP

   Name of Participant:

   TITLE: COMPARATIVE ANALYSIS BETWEEN RINGER'S LACTATE VS ACETATE CONTAINING BALANCED CRYSTALLOID SOLUTION (PLASMA LYTE-A) AS CARDIOPULMONARY BYPASS PRIME INFORMED CONSENT FORM Part-A: Patient Information Sheet We at PGIMER, Chandigarh are conducting research on Plasma Lyte-A as a CPB priming fluid. (Study title: COMPARATIVE ANALYSIS BETWEEN RINGER'S LACTATE VS ACETATE CONTAINING BALANCED CRYSTALLOID SOLUTION (PLASMA LYTE-A) AS CARDIOPULMONARY BYPASS PRIME). I am going to give you information and invite you to be part of this research. You will have full rights to decide whether or not you will participate in the research. Before you decide, you can talk to anyone (or your family physician) you feel comfortable with about the research. There may be some words that you do not understand. Please ask me to stop as we go through the information and I will take time to explain. If you have questions later, you can ask them of me, the study doctor or the staff).

   Purpose of the research Recent studies have demonstrated that better outcomes in terms of acidosis with the use of Plasma Lyte-A as Cardiopulmonary Bypass prime, being more physiological to plasma in composition. Thus, the present study compares the effects of Plasma Lyte-A as a priming flud with respect to ringer lactate.

   Type of Research Intervention This research will compare the possible effects of Plasma Lyte-A as CPB prime with respect to conventionally using ringer lactate in our institute.

   Participant selection We are inviting all patients of age >18 years undergoing Cardiopulmonary bypass for the coronary artery disease and heart valve surgeries in the department of Cardiothoracic and Vascular surgery, PGIMER to be a part of the study.

   Voluntary Participation Your participation in this research is entirely voluntary. It is your choice whether to participate or not. Whether you choose to participate or not, all the services you receive at this clinic will continue and nothing will change. If you choose not to participate in this research project, you will be offered the treatment that is routinely offered in this clinic/hospital for disease, and we will tell you more about it later. You may change your mind later and stop participating even if you agreed earlier.

   Procedures and Protocol This study involves analysis of arterial blood gases and lactic acid level assessment. It will be done a part of routine laboratory investigation for the patient undergoing cardiopulmonary bypass Reimbursements You will not be given any reimbursements to participate in the study. Confidentiality The information that we collect from this research project will be kept confidential. Information about you that will be collected during the research will be put away and no-one but the researchers will be able to see it. Any information about you will have a number on it instead of your name. Only the researchers will know what your number is and we will lock that information up with a lock and key. It will not be shared with or given to anyone except (name who will have access to the information, such as the investigators, Institutional Ethics committee, Data Safety Monitoring Board etc.). The data may be made accessible the concerned Regulatory Authorities and the Court of Law as and when required.

   Right to Refuse or Withdraw You do not have to take part in this research if you do not wish to do so. You may also stop participating in the research at any time you choose without having to give the reasons for doing so. It is your choice and all of your rights will still be respected.

   Alternatives to Participating If you do not wish to take part in the research, you will be provided with the established standard treatment available at PGIMER.

   Who to Contact In case of any queries during the study you can contact the investigators Dr. Harkant Singh+917087009554 Dr. Anand Kumar Mishra +7087009566 Dr. V.K. Arya +917087009531 Dr. DoniparthiPradeep +919493223593

   INFORMED CONSENT CERTIFICATE

   Study title: COMPARATIVE ANALYSIS BETWEEN RINGER'S LACTATE VS ACETATE CONTAINING BALANCED CRYSTALLOID SOLUTION (PLASMA LYTE-A) AS CARDIOPULMONARY BYPASS PRIME Name of the Institution: Post Graduate Institute of Medical Education and Research, Chandigarh.

   Documentation of the informed consent I have read the foregoing information, or it has been read to me. I have had the opportunity to ask questions about it and any questions that I have asked have been answered to my satisfaction. I consent voluntarily to participate as a participant in this research.

   Print Name of Participant__________________ Signature of Participant ___________________ Date ___________________________ Day/month/year If illiterate A literate witness must sign (if possible, this person should be selected by the participant and should have no connection to the research team). Participants who are illiterate should include their thumb-print as well.

   I have witnessed the accurate reading of the consent form to the potential participant, and the individual has had the opportunity to ask questions. I confirm that the individual has given consent freely.

   Print name of witness_____________________ Thumb print of participant Signature of witness ______________________ Date ________________________ Day/month/year

   Statement by the researcher/person taking consent

   I have accurately read out the information sheet to the potential participant, and to the best of my ability made sure that the participant understands the study and the purpose of the study.

   I confirm that the participant was given an opportunity to ask questions about the study, and all the questions asked by the participant have been answered correctly and to the best of my ability. I confirm that the individual has not been coerced into giving consent, and the consent has been given freely and voluntarily. A copy of this ICF has been provided to the participant.

   Print Name of Researcher/person taking the consent________________________

   Signature of Researcher /person taking the consent__________________________

   Date ___________________________ Day/month/year

   PATIENT PROFORMA

   Patient Name: Age/sex:

   Height: Weight: BSA:

   C.R.No: Admission No:

   Diagnosis:

   Date and time of surgery:

   Time of induction:

   Time of CPB start:

   Time of extubation:

   Parameter Pre operative Immediate post op After 12 hrs After 24hrs After 48 hrs Haemoglobin TLC Platelets Sodium Potassium Chloride Urea Creatinine Creatinine clearance Bilirubin Conjugated AST ALT ALP PT INR aPTT PTI

   Aortic cross clamp time:

   Duration of bypass:

   Additives added:

   ABG chart S.No Time pH pO2 pCO2 HCO3- S.B.E S. lactate Na+ K+ Cl-

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing heart valve surgeries under cardiopulmonary bypass
2. Patients undergoing coronary artery bypass graft surgeries for coronary artery disease under cardiopulmonary bypass

Exclusion Criteria:

1. Patients undergoing surgery for congenital heart diseases.
2. Patients of age less than 18 years.
3. Patients with liver dysfunction (Serum Bilirubin >1.2mg %).
4. Patients with renal dysfunction (Serum Creatinine >1.5mg %).
5. Patients with severe left ventricular dysfunction with ejection fraction <30%.
6. Patients undergoing cardiac surgeries in emergency conditions.
7. Patients undergoing CABG along with heart valve replacement or repair.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-02-10; Primary Completion 2017-09 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Change in Serum Lactate | Before induction, five minutes after CPB,five minutes after the termination of CPB, half an hour stay in the ICU soon after the patient is shifted from completion of surgery, before the patient is extubated
  Arterial blood gas analysis at before induction, five minutes after CPB, at the end of the termination of CPB, half an hour stay in the ICU soon after the patient is shifted from completion of surgery, before the patient is extubated

SECONDARY OUTCOMES:
Serum urea | Immediate post op, 12 hours, 24 hours and 48 hours after surgery
Serum creatinine | Immediate post op, 12 hours, 24 hours and 48 hours after surgery
Creatinine clearance | Immediate post op, 12 hours, 24 hours and 48 hours after surgery
Serum electrolytes | Immediate post op, 12 hours, 24 hours and 48 hours after surgery

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Hett DA, Smith DC. A survey of priming solutions used for cardiopulmonary bypass. Perfusion. 1994 Jan;9(1):19-22. doi: 10.1177/026765919400900104. PMID 8161863
- [Result] Gu YJ, Boonstra PW. Selection of priming solutions for cardiopulmonary bypass in adults. Multimed Man Cardiothorac Surg. 2006 Jan 1;2006(109):mmcts.2005.001198. doi: 10.1510/mmcts.2005.001198. PMID 24415398
- [Result] Morgan TJ, Power G, Venkatesh B, Jones MA. Acid-base effects of a bicarbonate-balanced priming fluid during cardiopulmonary bypass: comparison with Plasma-Lyte 148. A randomised single-blinded study. Anaesth Intensive Care. 2008 Nov;36(6):822-9. doi: 10.1177/0310057X0803600611. PMID 19115651
- [Result] Lang W, Zander R. Prediction of dilutional acidosis based on the revised classical dilution concept for bicarbonate. J Appl Physiol (1985). 2005 Jan;98(1):62-71. doi: 10.1152/japplphysiol.00292.2004. PMID 15591303
- [Result] Emmett M, Narins RG. Clinical use of the anion gap. Medicine (Baltimore). 1977 Jan;56(1):38-54. PMID 401925
- [Result] De Jonghe B, Cheval C, Misset B, Timsit JF, Garrouste M, Montuclard L, Carlet J. Relationship between blood lactate and early hepatic dysfunction in acute circulatory failure. J Crit Care. 1999 Mar;14(1):7-11. doi: 10.1016/s0883-9441(99)90002-3. PMID 10102718
- [Result] Lilley A. The selection of priming fluids for cardiopulmonary bypass in the UK and Ireland. Perfusion. 2002 Sep;17(5):315-9. doi: 10.1191/0267659102pf538oa. PMID 12243433
- [Result] Liskaser FJ, Bellomo R, Hayhoe M, Story D, Poustie S, Smith B, Letis A, Bennett M. Role of pump prime in the etiology and pathogenesis of cardiopulmonary bypass-associated acidosis. Anesthesiology. 2000 Nov;93(5):1170-3. doi: 10.1097/00000542-200011000-00006. PMID 11046201
- [Result] Alston RP, Theodosiou C, Sanger K. Changing the priming solution from Ringer's to Hartmann's solution is associated with less metabolic acidosis during cardiopulmonary bypass. Perfusion. 2007 Nov;22(6):385-9. doi: 10.1177/0267659108089142. PMID 18666740
- [Result] Murray DM, Olhsson V, Fraser JI. Defining acidosis in postoperative cardiac patients using Stewart's method of strong ion difference. Pediatr Crit Care Med. 2004 May;5(3):240-5. doi: 10.1097/01.pcc.0000112367.50051.3b. PMID 15115561